CLINICAL TRIAL: NCT04355650
Title: Clinical Pilot of Augmented Human Intelligence in Major Depressive Disorder (AHI/Depression Pilot)
Brief Title: Augmented Human Intelligence in Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William V. Bobo, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-005341
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical decision tool (Experimental): Launch of clinical decision support tool at baseline visit with study clinician.
  Interventions: Other: Clinical decision support tool

INTERVENTIONS:
Other: Clinical decision support tool — Adults (aged 18-64 years) who meet DSM-5 diagnostic criteria for non-psychotic unipolar major depressive disorder (MDD) and meet study eligibility criteria will receive 8 weeks of open-label treatment with an SSRI or SNRI antidepressant. Depressive symptoms will be assessed using the subject- and clinician-rated versions of the 16-items QIDS scale (QIDS-SR and QIDS-CR) and the 17-item HAMD at baseline, week 2 (via telephone), week 4, and week 8; with an additional phone contact at week 24. The QIDS scale scores at 2- and 4-weeks will be entered into the AHI-based clinical decision support tool, and the outcome predicted by the tool (e.g., the predicted eventual treatment outcome at 8 weeks) will be recorded. Clinicians and patients will be blinded to the clinical decision support tool prediction of outcome provided at the 2- and 4 weeks.

SUMMARY:
Researchers are testing whether a computer program (called a clinical decision support tool) can help clinicians predict how a patient with depression will respond to antidepressant medication.

ELIGIBILITY:
Recruitment by invitation only

Inclusion Criteria:

* Outpatients with nonpsychotic MDD. Outpatient status assumes that the subject is not psychiatrically hospitalized or in an active suicidal crisis requiring hospitalization.
* A total score of >10 on the QIDS-CR and on the QIDS-SR (equivalent to a HAMD17 score of 13 [ids-qids.org, accessed on April 12, 2019]) given that when medication exceeds the effect of placebo in primary care, participants have a 17-item HAMD score >12. We added 2 HAMD points to take into account the possibility of measurement error. This is a very similar approach taken to the successful recruitment of subjects into the PGRN-AMPS trial.
* Antidepressant treatment is deemed appropriate by the study clinician.
* Adults who are between 18-64 years of age.
* Ability to provide informed consent
* Ability to understand English

Exclusion Criteria:

* A medical contraindication that precludes SSRI or SNRI treatment.
* Presence of a general medical condition that, in the opinion of this study clinician, is the cause of their depressive symptoms, will be exclusionary.
* People with treatment-resistant depression will be excluded from participating. For this study, treatment resistance will be defined as failure to respond to two or more adequate therapeutic trials of SSRIs and at least on SNRI therapeutic trial (sufficient antidepressant dose, for 6 weeks or longer) during the current depressive episode. Failure to tolerate a therapeutic trial of a given medication (resulting in discontinuation due to adverse effects) will not be counted as exclusionary. Persons who have failed to respond to two or more adequately designed and executed therapeutic trials of SSRIs but have no history of least one failure to respond to SNRI treatment during the current depressive episode will be eligible to receive treatment with an SNRI in this study.
* Diagnosis of schizophrenia, schizoaffective disorder, bipolar I or II disorder, or bipolar disorder NOS (including other specified or other unspecified bipolar disorders) or a primary psychiatric condition that requires a different initial treatment than an antidepressant.
* Currently taking an antidepressant medication with subtherapeutic results in terms of antidepressive efficacy and unwilling to undergo a medication taper and discontinuation prior to initiation of a study drug from this protocol. The subject will be closely monitored by the study clinician during the medication taper and discontinuation phase. The design of the medication taper will be at the discretion of the study clinician. Subjects who cannot be safely tapered from their medication or who experience adverse effects during the taper that make further tapering infeasible will be excluded from the study.
* Use of antidepressant medication primarily for management of nicotine dependence, chronic pain, migraine prophylaxis or other diagnoses.
* Active substance use disorder. Persons in sustained full remission (> 12 months) and a negative urine drug of abuse screen at the screening visit will be considered eligible. Note: An additional urine drug screen will not be necessary for individuals with a negative urine drug screen documented in the medical record where the date of testing occurred within 12 weeks (84 days) of the screening/baseline study visit. However, study clinicians can still obtain a urine drug screen based on their clinical judgement even in participants with a negative drug screen within the 12 weeks preceding the screening/baseline study visit.
* Trazodone, melatonin, low-dose quetiapine (<100 mg QHS), z-drugs (zolpidem, zopiclone, eszopiclone, etc.), ramelteon, and diphenhydramine may be used as rescue medications for insomnia. Benzodiazepines may be used for treatment of anxiety, and atomoxetine may be used for the treatment of attention deficit disorder. Study subjects currently on antipsychotic medications (e.g., typical and atypical antipsychotic drugs, other than low-dose quetiapine for insomnia) and mood stabilizing agents (e.g., lithium, carbamazepine, valproate, lamotrigine) are not eligible for the study
* Pregnant subjects and those who are currently breastfeeding and who plan to continue breastfeeding will be excluded.
* Persons currently undergoing ECT, TMS or DBS as acute series or for maintenance.
* Patients currently psychiatrically hospitalized or in an active suicidal crisis requiring hospitalization in the opinion of the study clinician.
* Individuals whose total QIDS-CR and total QIDS-SR scores are 10 or higher at the screening visit but decrease (improve) to total scores less than 10 on either the QIDS-CR or QIDS-SR at the baseline visit

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Observed clinical outcomes compared to predicted outcome at 2 week follow up | Baseline to 2 week visit
  Evaluate the degree of statistical concordance between observed clinical outcomes (non-response/remission) after 8 weeks of treatment and the outcomes predicted by an AHI-based clinical decision support tool after 2 weeks of follow up (i.e., concordance between 2-week predicted outcome and 8-week observed outcome), as assessed using the QIDS-SR and QIDS-CR, in adults with DSM-5-defined MDD who receive prospective treatment with an SSRI or SNRI antidepressant.

SECONDARY OUTCOMES:
Observed clinical outcomes compared to predicted outcome at 4 week follow up | Baseline to 4 week visit
  Evaluate the degree of statistical concordance between observed clinical outcomes (non-response/remission) after 8 weeks of treatment and the outcomes predicted by an AHI-based clinical decision support tool after 4 weeks of follow up (i.e., concordance between 4-week predicted outcome and 8-week observed outcome), as assessed using the QIDS-SR and QIDS-CR, in adults with DSM-5-defined MDD who receive prospective treatment with an SSRI or SNRI antidepressant.

CONTACTS AND LOCATIONS:
Overall Officials: William V Bobo, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (2):
  • Study Protocol (2019-07-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT04355650/Prot_000.pdf
  • Informed Consent Form (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04355650/ICF_001.pdf